CLINICAL TRIAL: NCT00005610
Title: Aerosolized GM-CSF in the Treatment of Metastatic Melanoma to the Lung
Brief Title: Study of Aerosolized Sargramostim in Treating Patients With Melanoma Metastatic to the Lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N9975; CDR0000067739 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-05-02; First posted 2004-02-12 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Melanoma (Skin); Metastatic Cancer
Keywords: stage IV melanoma; recurrent melanoma; lung metastases
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sargramostim (Experimental): Patients receive aerosolized sargramostim (GM-CSF) over 10-15 minutes twice daily for 7 days. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline and prior to course 5.
  Patients are followed every 2 months for at least 1.5 years.
  Interventions: Biological: sargramostim

INTERVENTIONS:
Biological: sargramostim

SUMMARY:
RATIONALE: Colony-stimulating factors, such as sargramostim, may help the body's immune system to kill cancer cells. Giving sargramostim in different ways may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of sargramostim given as a breathing treatment for treating patients who have melanoma that is metastatic to the lung.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the therapeutic effects of aerosolized sargramostim (GM-CSF) in terms of progression free survival at 2 months and median survival rate in patients with metastatic melanoma to the lung. II. Determine the immunomodulatory effects of this treatment regimen in this patient population. III. Assess the quality of life in terms of physical and personal concerns of these patients treated with this regimen.

OUTLINE: Patients receive aerosolized sargramostim (GM-CSF) over 10-15 minutes twice daily for 7 days. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline and prior to course 5. Patients are followed every 2 months for at least 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed melanoma with radiographic evidence of prior or active involvement of the lung or pleura Measurable disease At least one lesion with at least one dimension in diameter of at least 10 mm on CT scan or MRI No non-measurable disease including the following: Bone lesions Leptomeningeal disease Ascites Pleural or pericardial effusion Inflammatory breast disease Lymphangitis cutis or pulmonis Unconfirmed abdominal masses not followed by imaging Cystic lesions

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,000/mm3 Platelet count at least 75,000/mm3 Hemoglobin at least 8.0 g/dL Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) AST no greater than 3 times ULN Renal: Creatinine no greater than 2.5 times ULN Cardiovascular: No New York Heart Association class III or IV heart disease Other: No uncontrolled infection Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 2 weeks since prior biologic or immunotherapy No other concurrent biologic or immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) No concurrent chemotherapy Endocrine therapy: At least 2 weeks since prior corticosteroids No concurrent systemic glucocorticosteroids Radiotherapy: At least 2 weeks since prior radiotherapy No concurrent radiotherapy Surgery: Not specified Other: No concurrent immunosuppressants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2000-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2 months
Median survival | Up to 1.5 years

SECONDARY OUTCOMES:
Quality of life | Up to 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, MD, PhD, Study Chair — Mayo Clinic
Locations (18):
- United States (18):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota